CLINICAL TRIAL: NCT05383287
Title: Characteristics, Phenotypes, and TRAITS of Heart Failure With Preserved Ejection Fraction (TRAITS-HFpEF)
Acronym: TRAITS-HFpEF
Status: Recruiting | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016CD012
Record Dates: First submitted 2022-04-25; First posted 2022-05-20 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFpEF)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — With the patient's consent, a blood sample of approximately 10mL may be donated for biobanking, allowing measurement of yet to be identified biomarkers including serum, plasma and DNA analysis. As technology is continually advancing it is not possible to comprehensively list analysis methods that may be applied to samples in the future, but it is expected that multiple types of analyses will be performed on the donated samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF), a certain type of heart failure, occurs when the heart doesn't pump blood around the body properly. It can cause breathlessness, tiredness, and swollen feet or ankles. It is not clear why people develop HFpEF and treatment options are very limited.

TRAITS-HFpEF is a study that aims to understand why people develop HFpEF, identify new tests and treatments, and gain information on the life expectancy of people living with this condition. It will do this by routinely collecting information on people attending a specialised outpatient HFpEF clinic.

DETAILED DESCRIPTION:
HFpEF represents the single largest unmet need in cardiovascular medicine (Butler et al, 2014). The proportion of patients with HFpEF ranges from 22 to 73% of all heart failure patients across all clinical settings, including primary care, hospital care and hospital admission (Ponikowski et al, 2016).

Treatment options in HFpEF are very limited, and several clinical trials have demonstrated neutral results when assessing survival benefit from medical therapy. A common theme for this is the heterogeneity that exists in the HFpEF patient population and non-targeted therapy is inadequate for this diverse population. Patients need to be characterised according to their clinical phenotypes and underlying biological mechanisms in order to provide targeted patient-specific treatment. (Shah et al, 2016)

TRAITS-HFpEF is an observational cohort study that aims to assess the epidemiology, and the association of clinical variables and outcomes of patients with HFpEF. A dedicated specialist HFpEF clinic provides the opportunity to recruit and collect data on a large cohort of patients that can provide insights into different HFpEF phenotypes and their associations and outcomes. This can help direct future research and delivery of specialist care.

All patients attending the HFpEF clinic at Manchester University NHS Foundation Trust (MFT) will be approached. The expectation is to recruit approximately 1,250 patients over a 5-year period. With the patients consent, a blood sample of approximately 10mL will be taken for biobanking to allow measurement of yet to be identified biomarkers, including plasma and DNA. This will be optional for patients. All clinical variables will be documented at the time of the recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the HFpEF clinic at MFT.

Exclusion Criteria:

* Age < 18 years
* Imprisonment
* Inability to provide full written or verbal informed consent in English

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All individuals will be considered for inclusion in this study regardless of age, disability, gender reassignment, marriage and civil partnership, pregnancy and maternity, race, religion and belief, sex, and sexual orientation except where the study inclusion and exclusion criteria explicitly state otherwise.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Composite of all cause mortality and hospitalisation for heart failure | 7.5 years

SECONDARY OUTCOMES:
All cause mortality | 7.5 years
Hospitalisation for heart failure | 7.5 years
Identification of HFpEF phenotypes | 7.5 years
  Machine Learning analysis will be implemented to assess relationships between multiple clinical variables and the aforementioned outcome measures to identify novel HFpEF phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Miller, MBChB, MRCP, Principal Investigator — Manchester University NHS FT
Locations (1):
- Manchester University NHS Foundation trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Participants will be asked to provide consent for pseudonymised study data, including, for example, individual patient-level data, scans and any other data collected as part of the study, to be shared for research purposes with investigators or organisations, including independent commercial organisations ('industry'), in the United Kingdom or overseas, including outside of the European Economic Area and in the United States of America. Participant personal details such as name, address, date of birth, contact details will not be shared.
Time Frame: Within the life time of the study
Access Criteria: Release of data or samples to investigators or organisations requesting access, whether they reside within or outside the UK, will be covered by Data and/or Material Transfer Agreements. The Agreements are legally binding documents that will regulate the use of data and/or samples to ensure that standards are maintained.

REFERENCES:
- [Background] Butler J, Fonarow GC, Zile MR, Lam CS, Roessig L, Schelbert EB, Shah SJ, Ahmed A, Bonow RO, Cleland JG, Cody RJ, Chioncel O, Collins SP, Dunnmon P, Filippatos G, Lefkowitz MP, Marti CN, McMurray JJ, Misselwitz F, Nodari S, O'Connor C, Pfeffer MA, Pieske B, Pitt B, Rosano G, Sabbah HN, Senni M, Solomon SD, Stockbridge N, Teerlink JR, Georgiopoulou VV, Gheorghiade M. Developing therapies for heart failure with preserved ejection fraction: current state and future directions. JACC Heart Fail. 2014 Apr;2(2):97-112. doi: 10.1016/j.jchf.2013.10.006. PMID 24720916
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191
- [Background] Shah SJ, Kitzman DW, Borlaug BA, van Heerebeek L, Zile MR, Kass DA, Paulus WJ. Phenotype-Specific Treatment of Heart Failure With Preserved Ejection Fraction: A Multiorgan Roadmap. Circulation. 2016 Jul 5;134(1):73-90. doi: 10.1161/CIRCULATIONAHA.116.021884. PMID 27358439